CLINICAL TRIAL: NCT03542383
Title: Treatment of Memory Disorders in Gulf War Illness With High Definition Transcranial Direct Cortical Stimulation
Acronym: GWI HDtDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, John Hart, Jr., Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-64; CDMRP-GW150060 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2018-05-07; First posted 2018-05-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Memory Disorders; Word Finding Difficulty
Keywords: Gulf War Illness; Memory; Word Finding; High Definition Transcranial Direct Current Stimulation; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Memory Disorders; Anomia

STUDY DESIGN:
Intervention Model Description: Participants with Gulf War Illness and word finding difficulty will be randomly assigned to either receive active tDCS or sham.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The assessors, tDCS administrators, and participants are masked to group assignment. Active and sham tDCS parameters are set up at each session by an experimenter who does not have contact with the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active HD tDCS (Active Comparator): Administer 10 20-minute sessions of 1 mA anodal High Definition Transcranial Direct Current Stimulation to the preSMA region over a two week period.
  Interventions: Device: High Definition Transcranial Direct Current Stimulation
- Sham HD tDCS (Sham Comparator): Administer 10 20-minute sessions of sham High Definition Transcranial Direct Current Stimulation to the preSMA region over a two week period.
  Interventions: Device: Sham High Definition Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: High Definition Transcranial Direct Current Stimulation — Administer 1 ma anodal HD tDCS over the preSMA for 20 minutes a session for 10 sessions over a two week period
  Arms: Active HD tDCS
Device: Sham High Definition Transcranial Direct Current Stimulation — Administer sham HD tDCS over the preSMA for 20 minutes a session for 10 sessions over a two week period
  Arms: Sham HD tDCS

SUMMARY:
A debilitating and common symptom in Gulf War Illnesses (GWI) is the inability to retrieve words. This affects one's conversations, ability to fluidly exchange information verbally and retrieve information from memory. The investigators have discovered 3 brain regions - the PreSupplementary Motor Area (preSMA), caudate nucleus, and the thalamus - that are essential for word retrieval. They have also detected abnormal EEG signals related to these regions in GWI patients who have problems retrieving words.

The investigators have used their model of verbal retrieval to design a noninvasive, nonpharmacological treatment that uses High Definition transcranial Direct Current Stimulation (HD tDCS). Using HD tDCS, they deliver small amounts of electric current to areas of the head to stimulate specific brain regions. The objective is to determine if delivery of HD tDCS over the preSMA will improve performance in GWI veterans with a verbal retrieval deficit. The investigators will administer pre-treatment tests of verbal retrieval measures while recording brain electrical activity. They will then administer 10 sessions of HD tDCS over the preSMA (20 minutes a session) in half the veterans. The other half will go through the same procedures, except the current will not be turned on (called the sham condition). The investigators will then compare performance between the "active" and sham group and assess if the treatment had a significant effect on performing verbal retrieval tasks and if there is a change in the ERP markers to account for how the treatment worked. If the treatment is found to be effective it will be offered to those in the sham group at the study's end.

The investigators predict this treatment regimen will lead to positive effects on a person's daily functions, especially improved conversational abilities, with few, if any, side effects. They hope to outline the standard procedures for physicians to perform the treatment by creating a manual on how to apply the treatment in a clinical setting so that it will be quickly available to use in multiple sites if the proposed study demonstrates that it is efficacious. This treatment can be made widely available for Warrior Transition Units, military clinics, and VA medical centers. In addition, if successful, this could potentially lead to development of other targets of stimulation to improve other cognitive deficits in GWI, and help alleviate verbal fluency deficits associated with other disorders.

DETAILED DESCRIPTION:
The objective of this proposal is to identify patients with GWI who have a verbal retrieval deficit and determine if delivery of HD tDCS over the PreSupplementary Motor Area of the brain (preSMA) will improve performance in verbal retrieval-related tasks.

Key cognitive symptom described by patients with GWI extends from a disruption in the cognitive process of verbal retrieval. This is manifested in a variety of dysfunctions including word retrieval deficits, verbal fluency disruption and potentially verbal episodic memory. The investigators have delineated a circuit of verbal retrieval using functional neuroimaging and electrophysiology measures in normal controls and in patient populations showing that a circuit of the preSMA-caudate nucleus-thalamus is essential for effective retrieval of verbal information. This model has generated specific ERP neural markers of successful verbal retrieval and we have studied GWI patients with dysfunction in these ERP and functional MRI markers.

In addition, patients with MS and TBI have been treated by the investigators for similar verbal retrieval deficits as those with GWI by using the technique of High Definition transcranial Direct Current Stimulation (HD tDCS) over the preSMA region to strengthen the connections of this retrieval circuit.

The investigators hypothesize that application of 1 ma anodal HD tDCS over the preSMA for 20 minutes a session for 10 sessions over a two week period will lead to improvement in verbal retrieval that will be detectable in both performance measures of verbal retrieval tasks and in ERP markers of verbal retrieval processing. The objective is to determine if 10 sessions of 1 ma anodal HD tDCS to the preSMA for 20 minutes a session are an effective treatment for verbal retrieval deficits in GWI.

The goal of this proposal is to entrain the verbal retrieval circuit using HD tDCS to target the preSMA in order to improve retrieval in impaired GWI patients, using behavioral and electrophysiological markers to assess outcomes. After identifying GWI patients with retrieval deficits using standard neuropsychological measures, the following aims will be addressed:

Aim 1. Administer 10 20-minute sessions of either 1 mA high definition tDCS or sham to the preSMA region.

Subtypes of Gulf War Illness patients have been shown to have dysfunction that disrupts the above-described retrieval circuit. Transcranial DCS targeted to the preSMA has been shown in preliminary studies in other diseased populations to result in improved performance in tasks that engage this circuit by purportedly strengthening potentially weak connections within the preSMA-caudate-thalamus circuit for verbal retrieval.

Hypothesis #1:HD tDCS to the preSMA will produce long-term modulation of the basal state of the preSMA-caudate-thalamic-cortical retrieval circuit.

Aim 2. Assess neuropsychological and electrophysiological (ERP) markers of verbal retrieval following tDCS therapy. Long-term modulation of the preSMA-caudate-thalamic-cortical retrieval circuit, via tDCS to the preSMA region, will alter the neurophysiological properties of the circuit due to modulation of the readiness of the retrieval circuit. This will result in changes in neural markers as follows:

Hypothesis #2a: Neuropsychological measures of verbal retrieval that were impaired at baseline will be improved to expected premorbid levels of functioning for the treated individuals.

Hypothesis #2b: Patients with impairments in making a correct retrieval will exhibit both high false negative errors and false positive errors compared to norms and a decreased 750-ms ERP amplitude difference between retrievals and nonretrievals on the SORT task. The investigators hypothesize that after HD tDCS treatment, these patients will improve performance and/or have an increase in amplitude difference in the ERP between retrievals and nonretrievals.

Hypothesis #2c: An increase in false negative errors and a decreased "Go" P3 ERP response on the Semantic Selection Tasks is indicative of an impaired ability to select a correct memory for retrieval. Conversely, there will be increased false positive errors and a decreased "NoGo" P3 ERP on the Semantic Selection Tasks if a patient cannot inhibit an incorrect memory. The investigators hypothesize that following HD tDCS therapy, there will be a normalization of the patient's behavior (reduced errors, improved RTs) and/or ERP responses (increased P3 amplitudes for Go and/or NoGo trials) due to modulation of the retrieval circuit, with the changes based on the pre-treatment impaired retrieval function (selection and/or inhibition).

ELIGIBILITY:
Inclusion Criteria:

* US military veterans serving during the 1990-1991 GW and were deployed to the theater of operations in Southwest Asia (i.e., Iraq, Kuwait, and Saudi Arabia) who are capable of understanding and signing an informed consent document.
* between the ages of 18 and 50 years old DURING SERVICE in the Gulf War (born between 1940 and 1973).
* Any gender, race/ethnicity, and both enlisted and officer ranks will be included.
* English speakers because not all of the screening forms, questionnaires, and tests are available in languages other than English.
* right-handed

Exclusion Criteria:

* non-English speakers because not all of the screening forms, questionnaires, and tests are available in any language except English.
* a history of a neurological disorder, including dementia of any type, moderate to severe traumatic brain injury (TBI), brain tumors, present or past drug abuse, stroke, blood vessel abnormalities in the brain, Parkinson's disease, Huntington's disease, or multiple sclerosis. Traumatic brain injury will be screened by history.
* anyone cognitively or clinically incompetent to give informed consent.
* taking medications that interact with the tDCS effect including amphetamines, L-dopa, carbamazepine, sulpiride, pergolide, lorazepam, rivastigmine, dextromethorphan, D-cycloserine, flunarizine, ropinirole,or citalopram.
* cardiac pacemakers, implanted medication pumps of any sort, or a history of bad heart disease, and/or the presence of any metal objects in or near the head which cannot be safely removed for the duration of this study which could be affected by tDCS or affect the administration of tDCS.

Ages: 45 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Change in performance on the Controlled Oral Word Association Test (COWAT) | Phone screen, beginning of HD tDCS/sham treatment, after HDtDCS/sham (2 weeks), at 3 month follow-up and 6 month follow-up.
  The COWAT is a verbal fluency test that measures spontaneous production of words belonging to the same category or beginning with some designated letter.
Change in the performance on the California Verbal Learning Test (CVLT) | Beginning of HD tDCS/sham treatment, after HDtDCS/sham (2 weeks), at 3 month follow-up and 6 month follow-up
  The CVLT is a measure of episodic verbal learning and memory. The test does this by attempting to link memory deficits with impaired performance on specific tasks. It assesses encoding, recall and recognition in a single modality of item presentation (auditory-verbal).

SECONDARY OUTCOMES:
Change in the performance on the Semantic Object Retrieval Test (SORT) | Beginning of HD tDCS/sham treatment, after HDtDCS/sham (2 weeks), at 3 month follow-up and 6 month follow-up
  The SORT was developed for the assessment of semantic memory and subsequent name production, and has been shown to detect word retrieval deficits in other neurological diseases.
Change in the performance on the Semantic Selection Task | Beginning of HD tDCS/sham treatment, after HDtDCS/sham (2 weeks), at 3 month follow-up and 6 month follow-up
  This is a go/no-go task performed during EEG.
Change in the performance on the Event Related Potential (ERP) | Beginning of HD tDCS/sham treatment, after HDtDCS/sham (2 weeks), at 3 month follow-up and 6 month follow-up
  ERP is the measured brain response that is the direct result of a specific sensory, cognitive, or motor event. This provides a noninvasive means of evaluating brain functioning. ERPs are measured by electroencephalography (EEG).

CONTACTS AND LOCATIONS:
Overall Officials: John Hart, Jr, MD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- Callier Center for Communication Disorders at The University of Texas at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Any information shared with other researchers will be de-identified.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT03542383/Prot_SAP_000.pdf